CLINICAL TRIAL: NCT02188732
Title: Self-Management Training and Automated Telehealth to Improve SMI Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen J. Bartels, Professor of Psychiatry, of Community and Family Medicine, and of TDI, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11522753
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Depression
Keywords: Community Mental Health; Serious Mental Illness; Medical Comorbidity; Self-Management; Automated Telehealth; Early Mortality
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depression | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBHH+AT (Experimental): Community Based Health Home + Automated Telehealth (CBHH+AT):
  Community-Based Health Home (CBHH) PLUS Automated Telehealth: a wireless telehealth device programmed with psychiatric content corresponding to the primary psychiatric diagnosis, and medical content tailored to the primary medical diagnosis. Daily interactive sessions last 5-10 min. Branching logic tailors questions or feedback to the user's responses (e.g., if a participant endorses medication nonadherence, a question appears asking why medications were not taken). The device automatically provides specific instructions to participants demonstrating signs of high risk.
  Interventions: Behavioral: CBHH+AT; Behavioral: CBHH
- CBHH+SMT (Active Comparator): CBHH+SMT Community-Based Health Home (CBHH) PLUS Self-Management Training (SMT) of I-IMR
  I-IMR integrates psychiatric illness self-management with strategies for medical illness self-management . The psychiatric component includes psychoeducation about illness and treatment, cognitive behavioral approaches to increase medication adherence, training and relapse prevention, teaching coping skills to manage persistent symptoms, and social skills training. The medical illness component consists of an individually tailored curriculum focused on managing physical illnesses using parallel skills and strategies taught for psychiatric illness self-management, as well as a nurse health care manager to facilitate coordination of necessary preventive and ongoing health care. The I-IMR curriculum consists of 10 modules delivered by an I-IMR specialist through eight months of weekly sessions customized to the specific needs and disorders of each client.
  Interventions: Behavioral: CBHH+SMT; Behavioral: CBHH
- CBHH (Active Comparator): Community-based Health Home (CBHH): Each team has a staff-to-participant ratio of approximately 1:12, with each team serving approximately 120 participants with SMI using person-centered planning and recovery-oriented, flexible service models. Each team provides mobile outreach and includes a team leader; a peer counselor; a psychiatric nurse coordinator; a clinical care coordinator; specialists in substance abuse (dual diagnosis), community integration, rehabilitation, employment, and housing; and a medical nurse practitioner (MNP) and a health outreach worker (HOW)
  Interventions: Behavioral: CBHH

INTERVENTIONS:
Behavioral: CBHH+AT — Community Based Health Home + Automated Telehealth (CBHH+AT):
  Community-Based Health Home (CBHH) PLUS Automated Telehealth: a wireless telehealth device programmed with psychiatric content corresponding to the primary psychiatric diagnosis, and medical content tailored to the primary medical diagnosis. Daily interactive sessions last 5-10 min. Branching logic tailors questions or feedback to the user's responses (e.g., if a participant endorses medication nonadherence, a question appears asking why medications were not taken). The device automatically provides specific instructions to participants demonstrating signs of high risk.
  Other Names: Person and Family-Centered Health Home; Automated Telehealth; Health Buddy
  Arms: CBHH+AT
Behavioral: CBHH+SMT — Illness Management and Recovery (IMR) for psychiatric illness combines (1) psychoeducation, which improves knowledge about mental illness management, (2) behavioral tailoring, which improves medication adherence, (3) relapse prevention training, which decreases relapses and rehospitalizations, and (4) coping skills training, which reduces distress related to symptoms. Illness Management and Recovery (I-IMR) by adding chronic medical illness self-management to psychiatric illness self-management. For each psychiatric self-management skill module, there is a corresponding medical illness self-management training component using established methods in self-management of common chronic health conditions (e.g., diabetes, hypertension, congestive heart failure, chronic obstructive pulmonary disease, etc.).
  Other Names: Illness Self-management; Self-mangement support; Integrated Illness Self-management and Recovery
  Arms: CBHH+SMT
Behavioral: CBHH — Community-based Health Home (CBHH): Each team has a staff-to-participant ratio of approximately 1:12, with each team serving approximately 120 participants with SMI using person-centered planning and recovery-oriented, flexible service models. Each team provides mobile outreach and includes a team leader; a peer counselor; a psychiatric nurse coordinator; a clinical care coordinator; specialists in substance abuse (dual diagnosis), community integration, rehabilitation, employment, and housing; and a medical nurse practitioner (MNP) and a health outreach worker (HOW).
  Other Names: Patient centered health home; Behavioral health home; Chronic disease management

SUMMARY:
This randomized clinical trial (RCT) of 300 persons with serious mental illness (SMI) and medical comorbidity will evaluate outcomes for n=100 in a Community Based Health Home alone (CBHH), compared to n=100 also receiving Self-Management Training (CBHH+SMT), and n=100 also receiving Automated Telehealth (CBHH+AT). The investigators will test the following 3 hypotheses:

Hypothesis 1: CBHH+SMT and CBHH+AT compared to CBHH alone, will be associated with greater health self-management and greater mental health self-management.

Hypothesis 2: CBHH+SMT and CBHH+AT compared to CBHH alone, will be associated with greater reduction in risk of early mortality and (Exploratory E2) in psychiatric symptoms.

Hypothesis 3: CBHH+SMT and CBHH+AT compared to CBHH alone, will be associated with less acute service use and less acute service use costs.

DETAILED DESCRIPTION:
Efforts to reduce early mortality in persons with serious mental illness (SMI) have largely focused on providing integrated primary care in a "health home". Yet medical care alone accounts for a disproportionately small contribution to reductions in early morality in comparison to improving self-management and health behaviors. Illness self-management training (SMT) in the general population has been shown to improve health outcomes and lower costs associated with chronic health conditions by teaching and coaching individuals on monitoring symptoms, self-administering treatments, and improving health behaviors. More recently, the use of technologies such as Automated Telehealth (AT) has been shown to improve outcomes and potentially prevent expensive emergency room and acute hospitalizations in the general population by daily prompting of self-management and remote monitoring by a nurse who can pre-emptively intervene, guided by disease management algorithms. To the investigators knowledge, neither of these approaches has been empirically evaluated as an integrated component in a behavioral health home for persons with SMI. The investigators will conduct a randomized clinical trial (RCT) of 300 persons with SMI and medical comorbidity to evaluate outcomes for n=100 in a Community Based Health Home alone (CBHH), compared to n=100 also receiving Self-Management Training (CBHH+SMT), and n=100 also receiving Automated Telehealth (CBHH+AT). The investigators will test the following 3 hypotheses:

Primary H1: CBHH+SMT and CBHH+AT compared to CBHH alone, will be associated with greater health self-management (measured by the Self Rated Abilities for Health Practices Scale) and (Exploratory E1) greater mental health self-management (measured by the Illness Management and Recovery Scale) at 4, 8, 12, and 24-months. Primary H2: CBHH+SMT and CBHH+AT compared to CBHH alone, will be associated with greater reduction in risk of early mortality (as measured by the Avoidable Mortality Risk Index) and (Exploratory E2) in psychiatric symptoms (BPRS) at 4, 8, 12, and 24 months. Primary H3: CBHH+SMT and CBHH+AT compared to CBHH alone, will be associated with less acute service use (emergency room visits and hospitalizations) and (Exploratory E3) less acute service use costs at 4, 8, 12, and 24-months.

In order to differentiate CBHH+SMT and CBHH+AT if both are found to be effective, the investigators will evaluate the persistence of primary outcomes from intervention endpoint (at 12 months) to the final follow-up (at 24 months) and will calculate the additional incremental costs of implementing and providing SMT and AT. The investigators will also explore differences in subjective health (SF-12) and in individual cardiovascular risk factors (e.g., BMI, tobacco use, blood pressure, glucose, lipids), comparing CBHH+SMT, CBHH+AT, and CBHH alone. Finally, the investigators will explore hypothesized mechanisms of action (potential mediators) for the Aim 2 primary outcome of reduced risk of early mortality (i.e., improvement in health self-management) and for the Aim 3 primary outcome of less acute service use (i.e., medication adherence and number of nurse preemptive interventions).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older and enrolled in treatment for at least 3 months;
2. SMI as defined by (i) primary DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder; (ii) moderate impairment across multiple areas of psychosocial functioning, including social relationships, self-care, community/work activity, treatment self-management, and community living skills; (iii) GAF (Global Assessment of Functioning) score less than 61. The broad range of SMI are included primarily because findings will be more generalizable to routine mental health settings, but also because we included this group in our pilot studies;
3. Diagnosis of one of the following medical illnesses or health conditions: diabetes, heart disease, chronic obstructive pulmonary disease, chronic pain, hyperlipidemia, hypertension, obesity, tobacco dependence;
4. Voluntary informed consent for participation in the study by the participant or by the participant's legally designated guardian;
5. An expressed willingness to participate in self-management training or a telehealth program;
6. Ability to read the telehealth display in English.

Exclusion Criteria:

1. Currently residing in a nursing home or group home;
2. Terminal physical illness expected to result in the death of the study subject within 12-24 months; or
3. Primary diagnosis of dementia, co-morbid diagnosis of dementia, or significant cognitive impairment as indicated by a Mini Mental State Examination (MMSE)74 score <24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Health Self-management | Change from baseline at 4,8,12, and 24 months
  Self Rated Abilities for Health Practices Scale
Change in risk of early mortality | Change from baseline at 4,8,12, and 24 months
  Avoidable Mortality Risk Index
Change in acute service use | Change from baseline at 4,8,12, and 24 months
  emergency room visits and hospitalizations

SECONDARY OUTCOMES:
Change in mental health self-management | Change from baseline at 4,8,12, and 24 months
  Illness Management and Recovery Scale
Change in psychiatric symptom severity | Change from baseline at 4,8,12, and 24 months
  Brief Psychiatric Rating Scale
Change in acute care costs | Change from baseline at 12 and 24 months
  emergency room and hospitalization costs

OTHER OUTCOMES:
Change in Subjective Health Status | Change from baseline at 4,8,12, and 24 months
  SF-12
Change in Cardiovascular Risk Factors | Change from baseline at 4,8,12, and 24 months
  BMI, Tobacco Use, Blood Pressure, Glucose, Lipids

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bay Cove Human Services, Boston, Massachusetts
  - Vinfen, Cambridge, Massachusetts

REFERENCES:
- [Background] Bartels SJ, Pratt SI, Mueser KT, Naslund JA, Wolfe RS, Santos M, Xie H, Riera EG. Integrated IMR for psychiatric and general medical illness for adults aged 50 or older with serious mental illness. Psychiatr Serv. 2014 Mar 1;65(3):330-7. doi: 10.1176/appi.ps.201300023. PMID 24292559
- [Background] Pratt SI, Bartels SJ, Mueser KT, Naslund JA, Wolfe R, Pixley HS, Josephson L. Feasibility and effectiveness of an automated telehealth intervention to improve illness self-management in people with serious psychiatric and medical disorders. Psychiatr Rehabil J. 2013 Dec;36(4):297-305. doi: 10.1037/prj0000022. PMID 24320837